## Comparative Study Between the Outcome of Intra-articular Injection of Platelet Rich Plasma Versus Hyaluronic Acid in Arthroscopic Management of Temporomandibular Degenerative Joint Diseases: A Randomized Clinical Trial

NCT04936945

11/5/2023

Table 1: VAS means for pain of the studied groups

| | Group HA<br>(n=10) | P1 | Group PRP<br>(n=10) | P2 | P value |
|---|---|---|---|---|---|
| Pre (mean±SD) | 49±20.79 | | 49±21.32 | | 1.00 |
| 1-week PO | 28±14.76 | 0.004* | 30±14.14 | 0.027* | 0.761 |
| 3-weeks PO | 21±8.76 | <0.001* | 25±14.34 | 0.011* | 0.461 |
| 1-month PO | 16±9.66 | <0.001* | 20±14.91 | 0.005* | 0.486 |
| 2-months PO | 13±6.75 | <0.001* | 13±9.49 | <0.001* | 1.000 |
| 3-months PO | 12±7.89 | <0.001* | 7±4.83 | <0.001* | 0.105 |
| 4-months PO | 12±10.33 | <0.001* | 4±5.16 | <0.001* | 0.042* |
| 5-months PO | 14±13.5 | <0.001* | 3±4.83 | <0.001* | 0.026* |
| 6-months PO | 14±13.5 | <0.001* | 3±4.83 | <0.001* | 0.026* |

<sup>\*</sup> Significant: P value ≤ 0.05, P1: P value compared to pre in HA group, P2: P value compared to pre in PRP group.



Fig 1 VAS means for pain of the studied groups.

The mean values of maximum interincisal mouth opening (MIO) were statistically analyzed both intragroup and intergroup, there was statistically significant increase in MIO in all postoperative follow-up periods in comparison with preoperative in both HA group and PRP group.

Intergroup comparison found no statistically significant differences between HA group and PRP group through all follow-up visits

Table 2: maximum interincisal opening (MIO) measurements of the studied groups

| | Group HA<br>(n=10) | P1 | Group PRP<br>(n=10) | P2 | P value |
|---|---|---|---|---|---|
| Pre (mean±SD) | 23.1±6.71 | | 27.9±4.51 | | 0.08 |
| 1-week PO | 33.8±3.43 | <0.001* | 35.6±3.69 | <0.001* | 0.27 |
| 3-weeks PO | 36±4.4 | <0.001* | 36.7±4.92 | <0.001* | 0.74 |
| 1-month PO | 36.7±5.08 | <0.001* | 37.3±5.5 | <0.001* | 0.80 |
| 2-months PO | 36.7±5.08 | <0.001* | 37.6±5.21 | <0.001* | 0.70 |
| 3-months PO | 37.6±4.55 | <0.001* | 38.2±4.71 | <0.001* | 0.78 |
| 4-months PO | 37.1±4.41 | <0.001* | 38±4.29 | <0.001* | 0.65 |
| 5-months PO | 36.8±4.78 | <0.001* | 38.3±4.06 | <0.001* | 0.46 |
| 6-months PO | 36.9±4.95 | <0.001* | 38.5±4.33 | <0.001* | 0.45 |

<sup>\*</sup> Significant: P value ≤ .05, P1: P value compared to pre in HA group, P2: P value compared to pre in PRP group.



Fig2 maximum interincisal opening (MIO) measurements of the studied groups